CLINICAL TRIAL: NCT02212002
Title: Effect of Intrapartum Antibiotic Prophylaxis (IAP) on the Development of Neonatal Gut Microbiota
Brief Title: Effect of Intrapartum Antibiotic Prophylaxis (IAP) on the Development of the Neonatal Gut Microbiota.
Acronym: MICROBIOTA-SO
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-2014-MICROBIOTA; 12/2013/U/Oss (Other: Ethic Committee of St. Orsola-Malpighi University Hospital (Bologna, Italy))
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Microbiota
Keywords: Group B Streptococcus; Intrapartum Antibiotic Prophylaxis; term infants; vaginal delivery; gut microbiota; feeding; molecular analysis; real-time PCR

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Control group: infants born to GBS-negative mothers, who thus did not receive any antibiotic treatment before/at delivery.
- IAP: IAP group: infants born to GBS-positive mothers who have received adequate intrapartum antibiotic prophylaxis (IAP). According to the Institutional treatment protocol for GBS prophylaxis (derived from CDC guidelines), intravenous ampicillin is given every 4 hours until delivery (first dose 2 g, following doses 1 g each). IAP is considered adequate when the mother received at least two doses of ampicillin before delivery.
  Interventions: Drug: IAP

INTERVENTIONS:
Drug: IAP — maternal IAP, consisting of intravenous ampicillin given every 4 hours until delivery (first dose 2 g, following doses 1 g each).
  Groups: IAP

SUMMARY:
The colonization of the neonatal gastro-intestinal (GI) tract begins at birth and is influenced by several factors, such as mode of delivery, gestational age, maternal intestinal and vaginal microbiota, type of feeding, hospitalization after birth and use of antibiotics and probiotics.

Gut microbiota of term infants, vaginally delivered and exclusively breastfed, shows a low count of C. difficile and E. coli and a high number of Bifidobacteria and Lactobacilli, which positively influence the host's immunity processes; hence, is considered to be ideally healthy.

Group B Streptococcus (GBS) represents one of the most important causes of neonatal infections and sepsis. Infants vaginally delivered may acquire GBS during the birth process from maternal vagina, cervix or rectum, where it resides in 10-20% of pregnant women. In the last decade, the incidence of early-onset GBS sepsis is significantly reduced, due to the introduction of GBS universal screening during late pregnancy and consequent intrapartum antibiotic prophylaxis (IAP) in GBS-positive women.

The use of antibiotics in early life is shown to alter the commensal gut microbiota, thereby impairing the balance between health and disease later in life. The effect of IAP on bacterial colonization of the infant's gut, however, has not been largely investigated. The investigators have previously evaluated the effect of IAP in a relatively small sample of exclusively breast-fed term infants vaginally delivered by means of molecular techniques; at 7 days of life there were several differences in microbiota composition between infants IAP-exposed and not exposed.

This observational prospective study thus aims to evaluate these differences in further detail, expanding the initial sample to formula-fed term infants and following up infants until one month of age. By including formula-fed infants, the investigators additionally aim to evaluate the influence of feeding type on the neonatal microbiota composition.

DETAILED DESCRIPTION:
At birth, the neonatal gastro-intestinal (GI) tract is rapidly colonized by maternal and environmental bacteria; the first colonizers are generally aerobes and facultative anaerobes, followed by strict anaerobes (e.g. Bifidobacterium spp., Bacteroides spp., and Clostridium spp.). The composition of gut microbiota is influenced by several factors, such as mode of delivery, gestational age, maternal intestinal and vaginal microbiota, type of feeding, hospitalization after birth and use of antibiotics and probiotics.

Gut microbiota of term infants, vaginally delivered and exclusively breastfed, is considered to be ideally healthy, with a low count of C. difficile and E. coli and a high number of Bidifobacteria and Lactobacilli, which positively influence the host's health by activating immunocompetent cells in the GI tract, promoting the production of secretory IgA and increasing the bactericidal activity of neutrophils and cell-mediated immunity such as NK cell activity.

Group B Streptococcus (GBS) is one of the most important causes of neonatal infections and sepsis. Infants vaginally delivered may acquire GBS during the birth process from maternal vagina, cervix or rectum, where it resides in approximately 10-20% of pregnant women. Since the mid-90s, the incidence of early-onset GBS sepsis is significantly reduced, due to the introduction of GBS universal screening during late pregnancy and consequent intrapartum antibiotic prophylaxis (IAP) in GBS-positive women.

Recent data suggest that the use of antibiotics in early life could alter the commensal gut microbiota, thereby impairing the balance between health and disease later in life. The effect of IAP on bacterial colonization of the infant's gut has not been largely investigated. Moreover, currently available data on this issue largely derive from studies performed using culture-based techniques; however, accurate culture-based results are influenced by the selection of the correct media, temperature, oxygen content and time for growth, and for this reason as little as 10-50% of the entire gut bacteria are easily cultured. Molecular techniques, based on the amplification of the 16S ribosomal bacterial RNA gene to differentiate prokaryotic taxa, have been recently developed for the study of gut microbiota, thus enabling a more detailed characterization of bacterial communities than standard culture.

We have previously evaluated the effect of IAP in a relatively small sample of exclusively breast-fed term infants vaginally delivered by means of molecular techniques; at 7 days of life there were several differences in microbiota composition between infants IAP-exposed and not exposed.

The aim of the present paper is thus to evaluate these differences in further detail, expanding the initial sample and following up infants until one month of age. Influences of type of feeding on microbiota composition are also explored.

Healthy term infants, vaginally delivered, with birth weight adequate for gestational age, and whose mothers had been screened for GBS at 35-37 weeks gestation, are enrolled in the study.

Infants are excluded if:

* preterm or small/large for gestational age
* born by caesarean section
* the mother has received any antibiotic in the 4 weeks before delivery;
* maternal IAP is performed for reasons other than GBS positivity (i.e. prolonged rupture of membranes in GBS-negative women);
* maternal IAP is inadequate;
* maternal IAP is performed with antibiotics other than ampicillin, such as erythromycin;
* the infant has major congenital malformations;
* the infant develops signs of infection and/or received any antibiotic treatment after birth;
* the infant has any serious clinical conditions that contraindicated his/her participation in the study.

Infants are allocated into two groups according to maternal GBS status and IAP:

* IAP group: infants born to GBS-positive mothers who have received adequate IAP. According to the Institutional treatment protocol for GBS prophylaxis (derived from CDC guidelines), iv ampicillin is given every 4 hours until delivery (first dose 2 g, following doses 1 g each). IAP is considered adequate if the mother has received at least two doses of ampicillin before delivery.
* Control group: infants born to GBS-negative mothers, who do not receive any antibiotic treatment before/at delivery.

Written informed consent is obtained from each infant's parent/legal guardian when the infant is about to be discharged from the nursery (48-72 hours of life). Patients' characteristics, including gestational age, birth weight, gender, and Apgar score at 1' and 5' after birth, are summarized in a specific case report form.

Two faecal samples from each infant are collected during follow up visits at 7 and 30 days of life. At each visit, information on weight gain, clinical conditions, feeding, and on-going treatments (i.e. use of prebiotics, probiotics, antibiotics), are collected from the infants' parents.

After collection, faecal samples are put into numbered screw-capped sterile plastic containers and immediately frozen at -80 °C, until they are processed for bacterial DNA extraction.

Microbiological analyses are performed at the Department of Agricultural Sciences, University of Bologna. Investigators who perform the analyses are blind to group identity of the infants (IAP or control group).

Two hundred milligrams of faeces are used for bacterial DNA extraction using the QIAamp DNA Stool Mini Kit (QIAGEN, West Sussex, UK). Extracted DNA is stored at -80 °C. The purity and concentration of extracted DNA are determined by measuring the ratio of the absorbance at 260 and 280 nm (Infinite® 200 PRO NanoQuant, Tecan, Mannedorf, Switzerland).

Quantification of selected microbial groups (Lactobacillus spp., Bifidobacterium spp., Bacteroides fragilis) is performed with real-time PCR. Data obtained from amplification are transformed to obtain the number of bacterial cells per gram of faeces, expressed as log colony forming unit (CFU)/g.

The obtained data are analyzed using IBM SPSS Statistic version 20.0.0 (IBM Corporation, IBM Corporation Armonk, New York, United States). Baseline characteristics in the IAP and control groups are compared using the independent-samples Mann-Whitney U test for continuous variables and chi-square test for categorical variables. The influence of IAP on faecal bacterial count at 7 and 30 days of life will is evaluated using the independent-samples Mann-Whitney U test. A hierarchical multiple regression analysis is performed in order to estimate the effect of IAP on faecal bacterial count after controlling for type of infant feeding (coded as a binary categorical variable: exclusive breastfeeding vs. any formula feeding). A p value <0.05 is considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Term newborns (gestational age ≥ 37 weeks), vaginally delivered newborn
* birth weight adequate for gestational age
* mothers screened for GBS at 35-37 weeks gestation
* Obtained written parental consent.

Exclusion Criteria:

* Preterm or small/large for gestational age infants;
* Infants born by caesarean section;
* Infants admitted to the Neonatal Intensive Care Unit;
* Infants with major congenital malformations;
* Infants who received any antibiotic treatment after birth;
* Signs of infection and/or any serious clinical conditions that contraindicate the participation in the study;
* Infants whose mother had received any antibiotic in the 4 weeks before delivery;
* maternal IAP performed for reasons other than GBS positivity (i.e. prolonged rupture of membranes in GBS-negative women);
* inadequate maternal IAP;
* maternal IAP performed with antibiotics other than ampicillin, such as erythromycin

Max Age: 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: At least 60 infants (IAP group n=30, control group n=30), born at Sant'Orsola-Malpighi University Hospital and fulfilling the inclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Faecal bacterial count | One month
  Reduction in the faecal bacterial count (Bifidobacterium spp., Lactobacillus spp. and Bacteroides fragilis), assessed in term and vaginally delivered infants, in relation to IAP exposition.

CONTACTS AND LOCATIONS:
Locations (1):
- Nursery, S.Orsola-Malpighi Hospital, Bologna, Italy